CLINICAL TRIAL: NCT03918291
Title: Whole-body Vibration Training on Muscle Strength and Brain-derived Neurotrophic Factor Levels in Elderly Woman With Knee Osteoarthritis: a Randomized Clinical Trial Study.
Brief Title: Whole-body Vibration Training on Functional Performance of the Elderly With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1231-3069; 046.08 (Other: Federal University of Jequitinhonha and Mucuri Valleys)
Record Dates: First submitted 2019-04-10; First posted 2019-04-17 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis of Knee
Keywords: Muscle strength; Squat; Brain derived neurotrophic factor; Osteoarthritis of knee; Whole-body vibration; Elderly
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial in which the variables were assessed 24 h before and 24 h after a 12-week training program. For the allocation of participants, a 1:1 ratio randomization was performed.
Who Masked: Outcomes Assessor
Masking Description: The tests were performed by an experienced examiner who was blind to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addition of whole-body vibration to squat training (Experimental): The addition of whole-body vibration to squat training (for 12 weeks, 3x/week). The mechanical stimulation parameters of the vibration consisted of the following: frequency of 35 to 40 Hz, amplitude of 4 mm and acceleration that ranged from 2.78 to 3.26 G
  Interventions: Other: Addition of whole-body vibration to squat training
- Squat training (Other): Squatting exercises for 12 weeks, 3x/week
  Interventions: Other: Squat training

INTERVENTIONS:
Other: Addition of whole-body vibration to squat training
  Arms: Addition of whole-body vibration to squat training
Other: Squat training — squatting exercises for 12 weeks, 3x/week
  Arms: Squat training

SUMMARY:
The present study evaluated the effects of adding whole body vibration to squat training on the isometric quadriceps muscle strength, the plasma concentration of brain-derived neurotrophic factor at rest in elderly woman with osteoarthritis of the knee. The eligible patients were fifteen elderly women ≥ 60 years of age who had been diagnosed with osteoarthritis of the knee. The intervention consisted of uninterrupted squatting exercises for 12 weeks, a 3x/week. The exercise protocol was similar in both groups differed only in the presence of vibration.

DETAILED DESCRIPTION:
Ethical statement: This study was carried out in accordance with the recommendations of the ethical principles for research involving humans (Resolution 196-96 of the National Health Council of the Brazilian Ministry of Health) and Federal University of Jequitinhonha and Mucuri Valleys Ethics Committee. All subjects gave written informed consent in accordance with the Declaration of Helsinki. The protocol was approved by the Federal University of Jequitinhonha and Mucuri Valleys Ethics Committee (protocol No. 046.08).

Design: This is a randomized, controlled trial in which the variables were assessed 24 h before and 24 h after a 12-week training program. For the allocation of participants, a 1:1 ratio randomization was performed using opaque envelopes for allocation concealment. To minimize the chance of bias, The investigators used the following methods: a) opaque, sealed and serial-numbered envelopes; b) the envelopes were opened sequentially after the participant name and details were written on the envelope; c) the envelopes were kept in a locked and secure place. The allocation sequence was concealed from the researcher enrolling and assessing participants. Only one researcher performing the randomization was aware of the group assignment.

Subjects: The particpants were recruited through the physiotherapy clinic and through medical referrals. To participate in the study, participants were required to meet the following inclusion criteria: females older than 65 years of age; not using hormone replacement therapy; diagnosed with OA in at least one knee in accordance with of the American College of Rheumatology. The severity of the kOA was classified radiographically according to the Kellgren and Lawrence scale (grades 0-4, with 0 being normal and 4 representing severe OA). A Grade 2 classification (definite osteophytes and possible narrowing of joint space) was used as a cutoff to determine knee OA. Further inclusion criteria included the following: no recent knee injury; no walking aid requirement; and no rehabilitation procedures in the previous three months. Participants were excluded if they had any orthopedic, neurological, respiratory or acute cardiac diseases or if had any cognitive deficit as determined by the Mini-Mental State Examination.

Of the 125 elderly people screened for eligibility, 15 elderly women fulfilled the criteria, had blood sampling collected at rest (8:00 a.m.) and then participated in the IQMS test. Thereafter, the participants were allocated to one of two groups: 1) the vibration group, in which participants performed squat exercise training in association with WBV (VG; n=7); or 2) the exercise group, in which participants performed squat exercise training without vibration (EG; n=8).

Procedures: The clinical and demographic data were collected from the participants using an evaluation chart. Prior to the initiation of the 12-week intervention program, a blood sample was collected at 8:00 a.m. from the volunteers of all groups followed by the isometric quadriceps muscle strength (IQMS) evaluation. At 24 h after the intervention period, the volunteers of both groups were reassessed. These procedures were performed to avoid any circadian rhythm effects on hormonal status and the performance of IQMS. The tests were performed by an experienced examiner who was blind to the group allocation.

The intervention program consisted of performing squat exercise training with (VG) or without (EG) whole body vibration, three times a week on alternate days.

Warm-up: Prior to each training session, the participants warmed-up on a stationary cycle at 70% of the predicted maximum heart rate for each subject's age and were monitored using a Polar heart rate monitor (Polar F4, Kempele, Finland) for 10 minutes. Immediately afterwards, the participants of the VG group were placed in a position with their feet 28 cm apart (14 cm to the right and 14 cm to the left of the center of the vibration stimulus) and were ready to begin the squat exercises on the vibratory platform, while the participants of the EG group performed the same procedure without vibration.

Squat exercises: The intensity of squat exercise training was systematically augmented in the vibration and exercise groups over the training period by increasing the number of repetitions (6 x 20 seconds to 8 x 40 seconds) and reducing the resting time (40 to 25 seconds). During each exercise repetition, the examiner instructed the volunteer to perform 3 seconds of isometric flexion of the quadriceps at 60º and 3 seconds of isometric flexion of the quadriceps at 10º. The 60º angle was measured in each volunteer using a universal goniometer prior to initiating the exercise series, and a barrier was placed at the gluteal region to limit the degree of flexion of the knee. The participants of both groups were placed in position with their feet 28 cm apart.

Whole body vibration: For the participants in the VG group, a commercial model of a vibration platform was used (FitVibe, GymnaUniphy NV, Bilzen, Belgium). In this group, acceleration was also increased by varying the vibration frequency (35-40 Hz). The mechanical stimulation parameters of the vibration consisted of the following: frequency of 35 to 40 Hz, an amplitude of 4 mm and acceleration that ranged from 2.78 to 3.26 G. The platform provided a vertical sinusoidal vibration. Prior to initiating data collection, the platform acceleration values were verified using the Mega accelerometer (Acceleration Measuring Kit ZPP1-3D-147BC, Southampton, United Kingdom).

To measure acceleration on the horizontal and vertical axes, two accelerometers (Acceleration Measuring Kit ZPP1-3D-147BC, Southampton, United Kingdom) were fixed at a distance of 14 cm from the center of platform vibration. The signal was amplified electronically and was stored. This signal was obtained at a frequency of 1000 Hz and was sent for computer analysis. Each accelerometer was calibrated using two calibration points and applying zero and gravity, Earth's gravity is 1 G (9.81 m/s2). To obtain the true acceleration values of the platform, the values of Earth's gravity were subtracted along the vertical axis from the total signal received so that the acceleration of the platform would begin at 0 m/s2. The data were transferred to a computer using the Megawin software program, and the mean and maximum acceleration of each sample on each axis were analyzed using the Matlab software program. Each frequency used was measured over 60 seconds. In the pilot study, interexaminer reliability was found to be high, with a coefficient of variation of 1.05%.

The participants underwent training on the vibratory platform with barefoot to avoid any damping effect due to different footwear. In addition, a predetermined distance from the feet (14cm to the right and 14cm to the left of the vibration center of the platform) was set to ensure that each of the lower limbs received the same amount of vibration stimulus. Moreover, with the aim of maintaining control of the body's center of gravity behind the base of the support, the positioning of the spine, arms, and head and the type of squat (simulating the motion of sitting in a chair) were standardized.

Isometric quadriceps muscle strength (IQMS): The IQMS was evaluated by the maximal voluntary isometric contraction of knee extensors (MVIC) measured using the load cell. For this evaluation, the participant was positioned in a flexion-extension chair (Home Sport, Master Top model, Belo Horizonte, Brazil) and assumed a sitting posture with a straight trunk and the hips flexed at 90º. The limb to be tested was positioned at 60° of knee flexion (assessed individually by goniometry of the knee), and the resistance lever was positioned on the distal leg.

The load cell was properly calibrated and positioned near the leg extension perpendicular to the ground for signal acquisition during the isometric muscle strength tests (Miotec - Biomedical Equipment, Porto Alegre, Brazil). The load cell was connected to the software MIOTOOL 400 that transmitted the isometric muscle strength values to a computer. The MVIC test was performed for 6 seconds with 1 minute between sets and with repeating three sets per leg.

Before the test, the participants warmed up for 10 minutes on a stationary bicycle (Stone Fitness, 2001, Huntertown, United State), which stimulated the heart rate (HR) to 70% of the estimated maximum HR by age, as measured with the use of the Polar heart monitors (Polar F4, Kempele, Finland). This procedure was performed to reduce the risk of injury during testing.

The intra-class correlation coefficient (ICC) for IQMS was 0.98 (95% CI: 0.94-0.99).

Analysis of BDNF by ELISA: For plasma processing, 10-mL peripheral blood samples were collected from the antecubital vein using aseptic techniques and heparin as an anticoagulant. The blood was immediately centrifuged twice at 3,000 g for 10 min, and the plasma was kept frozen at -70º C until assayed. Plasma BDNF levels were measured in duplicate using ELISA kits for BDNF (BDNF DuoSet, R&D Systems) according to the manufacturer's instructions; the detection limit was 10 pg/mL.

ELIGIBILITY:
Inclusion Criteria:

* females older than 65 years of age
* not using hormone replacement therapy
* diagnosed with OA in at least one knee in accordance with of the American College of Rheumatology

Exclusion Criteria:

* no recent knee injury
* no walking aid requirement
* no rehabilitation procedures in the previous three months
* any orthopedic, neurological, respiratory or acute cardiac diseases
* any cognitive deficit as determined by the Mini-Mental State Examination

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10-28 (Actual); Primary Completion 2010-10-28 (Actual); Study Completion 2012-06-28 (Actual)

PRIMARY OUTCOMES:
Change in isometric quadriceps muscle strength | 24 hours before and 24 hours after a 12-week training program
  The maximal voluntary isometric contraction of knee extensors measured using the load cell

SECONDARY OUTCOMES:
Change in plasma concentration of neurotrophin 40/5000 Plasma neurotrophin concentration | 24 hours before and 24 hours after a 12-week training program
  Brain derived neurotrophic factor plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cristina R Lacerda, PhD, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simao AP, Mendonca VA, Avelar NCP, da Fonseca SF, Santos JM, de Oliveira ACC, Tossige-Gomes R, Ribeiro VGC, Neves CDC, Balthazar CH, Leite HR, Figueiredo PHS, Bernardo-Filho M, Lacerda ACR. Whole Body Vibration Training on Muscle Strength and Brain-Derived Neurotrophic Factor Levels in Elderly Woman With Knee Osteoarthritis: A Randomized Clinical Trial Study. Front Physiol. 2019 Jun 25;10:756. doi: 10.3389/fphys.2019.00756. eCollection 2019. PMID 31293437